CLINICAL TRIAL: NCT01175369
Title: School-Based Asthma Therapy: Stage 2 Effectiveness Study
Acronym: SBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Halcyon Hill Foundation (Other)
Responsible Party: Principal Investigator, Jill Halterman, Associate Professor of Pediatrics, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 12308; 1R01HL079954-01A1 (NIH); NCT00296998 (obsolete NCT alias)
Record Dates: First submitted 2010-06-23; First posted 2010-08-04 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2013-08

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Usual asthma care
- School-based Care (Experimental): The intervention includes directly observed administration of preventive medications in school and a home-based ETS reduction program (for those living with one or more smokers).
  Interventions: Behavioral: School-based Care

INTERVENTIONS:
Behavioral: School-based Care — The intervention includes directly observed administration of preventive medications in school and a home-based ETS reduction program (for those living with one or more smokers).
  Arms: School-based Care

SUMMARY:
Asthma is the most common chronic illness of childhood, and hospitalization rates are increasing. In the US, impoverished children and children from minority ethnic and racial backgrounds suffer disproportionately from asthma. While National Heart, Lung, and Blood Institute (NHLBI) guidelines recommend daily preventive medications for all children with mild persistent to severe persistent asthma, studies indicate that many children in the US who should receive preventive medications are not receiving them. The overall goal of this project is to target an ethnically diverse population of inner-city schoolchildren with asthma and explore a school-based program to reduce asthma morbidity. We hypothesize that children receiving a comprehensive school-based intervention will experience less asthma-related morbidity compared to children receiving usual care. Our comprehensive school-based intervention consists of both administration of recommended preventive asthma medications in school (with dose adjustments according to NHLBI guidelines) and an environmental tobacco smoke (ETS) reduction program in the home for smoke-exposed children. Our secondary hypothesis is that, among the subgroup of smoke-exposed children, those who receive the school-based intervention with ETS reduction will experience less asthma morbidity than those who receive usual care.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma
* Mild persistent to severe persistent asthma
* Ages 3-10 years
* Attending school in the Rochester City School District preschools or elementary schools
* Signed physician permission to enroll the child
* Parent or caregiver must consent to the intervention

Exclusion Criteria:

* Inability to speak and understand either English or Spanish
* No access to a working phone for follow-up surveys
* The family planning to leave the school district within fewer than 6 months
* The child having other significant medical conditions that could interfere with the assessment of asthma-related outcome measures
* children in foster care or other situations in which consent cannot be obtained from a guardian
* Current participation in other local asthma interventions

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 530 (Actual)
Dates: Start 2006-08; Primary Completion 2009-06 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill S. Halterman, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Halterman JS, Borrelli B, Fisher S, Szilagyi P, Yoos L. Improving care for urban children with asthma: design and methods of the School-Based Asthma Therapy (SBAT) trial. J Asthma. 2008 May;45(4):279-86. doi: 10.1080/02770900701854908. PMID 18446591
- [Background] Fagnano M, van Wijngaarden E, Connolly HV, Carno MA, Forbes-Jones E, Halterman JS. Sleep-disordered breathing and behaviors of inner-city children with asthma. Pediatrics. 2009 Jul;124(1):218-25. doi: 10.1542/peds.2008-2525. PMID 19564303
- [Background] Conn KM, Hernandez T, Puthoor P, Fagnano M, Halterman JS. Screen time use among urban children with asthma. Acad Pediatr. 2009 Jan-Feb;9(1):60-3. doi: 10.1016/j.acap.2008.10.001. PMID 19329093
- [Background] Halterman JS, Borrelli B, Tremblay P, Conn KM, Fagnano M, Montes G, Hernandez T. Screening for environmental tobacco smoke exposure among inner-city children with asthma. Pediatrics. 2008 Dec;122(6):1277-83. doi: 10.1542/peds.2008-0104. PMID 19047246
- [Background] Halterman JS, Borrelli B, Conn KM, Tremblay P, Blaakman S. Motivation to quit smoking among parents of urban children with asthma. Patient Educ Couns. 2010 May;79(2):152-5. doi: 10.1016/j.pec.2009.09.004. Epub 2009 Sep 30. PMID 19796913
- [Background] Shone LP, Conn KM, Sanders L, Halterman JS. The role of parent health literacy among urban children with persistent asthma. Patient Educ Couns. 2009 Jun;75(3):368-75. doi: 10.1016/j.pec.2009.01.004. Epub 2009 Feb 23. PMID 19233588
- [Background] Fagnano M, Conn KM, Halterman JS. Environmental tobacco smoke and behaviors of inner-city children with asthma. Ambul Pediatr. 2008 Sep-Oct;8(5):288-93. doi: 10.1016/j.ambp.2008.04.002. Epub 2008 May 12. PMID 18922501
- [Background] Fagnano M, Bayer AL, Isensee CA, Hernandez T, Halterman JS. Nocturnal asthma symptoms and poor sleep quality among urban school children with asthma. Acad Pediatr. 2011 Nov-Dec;11(6):493-9. doi: 10.1016/j.acap.2011.05.006. Epub 2011 Aug 3. PMID 21816697
- [Background] Fagnano M, Halterman JS, Conn KM, Shone LP. Health literacy and sources of health information for caregivers of urban children with asthma. Clin Pediatr (Phila). 2012 Mar;51(3):267-73. doi: 10.1177/0009922811421413. Epub 2011 Sep 12. PMID 21911409
- [Background] Blaakman S, Tremblay PJ, Halterman JS, Fagnano M, Borrelli B. Implementation of a community-based secondhand smoke reduction intervention for caregivers of urban children with asthma: process evaluation, successes and challenges. Health Educ Res. 2013 Feb;28(1):141-52. doi: 10.1093/her/cys070. Epub 2012 Jun 20. PMID 22717938
- [Background] Noyes K, Bajorska A, Fisher S, Sauer J, Fagnano M, Halterman JS. Cost-effectiveness of the School-Based Asthma Therapy (SBAT) program. Pediatrics. 2013 Mar;131(3):e709-17. doi: 10.1542/peds.2012-1883. Epub 2013 Feb 11. PMID 23400614
- [Background] Koehler AD, Fagnano M, Montes G, Halterman JS. Elevated burden for caregivers of children with persistent asthma and a developmental disability. Matern Child Health J. 2014 Nov;18(9):2080-8. doi: 10.1007/s10995-014-1455-6. PMID 24619226
- [Background] Evans KA, Halterman JS, Hopke PK, Fagnano M, Rich DQ. Increased ultrafine particles and carbon monoxide concentrations are associated with asthma exacerbation among urban children. Environ Res. 2014 Feb;129:11-9. doi: 10.1016/j.envres.2013.12.001. Epub 2014 Jan 11. PMID 24528997
- [Result] Halterman JS, Szilagyi PG, Fisher SG, Fagnano M, Tremblay P, Conn KM, Wang H, Borrelli B. Randomized controlled trial to improve care for urban children with asthma: results of the School-Based Asthma Therapy trial. Arch Pediatr Adolesc Med. 2011 Mar;165(3):262-8. doi: 10.1001/archpediatrics.2011.1. PMID 21383275

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | School-based Care
Started | 265 | 265
Completed | 263 | 260
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | School-based Care | Total
Number analyzed (Participants) | 265 | 265 | 530
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 265 | 265 | 530
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.2 (1.9) | 7.1 (2.0) | 7.1 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 104 | 222
  Male | 147 | 161 | 308
Region of Enrollment [Number; unit: participants]
  United States | 265 | 265 | 530

OUTCOME MEASURES:

1. Primary Outcome: Number of Symptom Free Days
Description: The primary outcome variable is the average number of symptom free days over 2 weeks assessed during peak asthma season (data collected during November, December, January and February during the school year).
Time Frame: Average Symptom Free Days, over 2 weeks, during peak asthma season (November-February)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Usual Care | School-based Care
Number analyzed (Participants) | 263 | 260
Days | 10.7 (3.1) | 11.6 (2.5)

2. Secondary Outcome: Cotinine Level
Description: To test the effectiveness of the environmental tobacco smoke (ETS) reduction portion of the study, we will compare baseline cotinine values to 2 month (for smoke exposed participants) and final follow-up assessments (for all participants).
Time Frame: 2 month and approximately 9 month (end of school year) follow-up assessments
Reporting Status: Not Posted

3. Secondary Outcome: Cost Effectiveness of the Intervention
Description: Cost-effectiveness will examine the net program costs to the number of symptom-free days gained. Benefits will be described as the net difference in medical and productivity costs between children in the treatment and control groups.
Time Frame: approximately 9 months (length of school year)
Reporting Status: Not Posted

4. Secondary Outcome: Additional Asthma Morbidity Outcomes
Description: We will look at additional asthma morbidity outcomes including symptom nights, days needing rescue medications, functional severity, days absent from school, and quality of life.
Time Frame: 1-9 months (Monthly Follow-up assessments)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Usual Care | School-based Care
Serious Adverse Events (participants affected / at risk) | 0/265 | 0/265
Other Adverse Events (participants affected / at risk) | 0/265 | 0/265

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No